CLINICAL TRIAL: NCT02492243
Title: Continuous Rhythm Monitoring in Patients After Acute Myocardial infaRction and pREServed Left venTricle Ejection Fraction
Brief Title: Continuous Rhythm Monitoring in Patients After Acute Myocardial infaRction andpREServed Lef venTricle Ejection Fraction (ARREST)
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Meshalkin Research Institute of Pathology of Circulation (Network)
Collaborators: Medtronic Cardiac Rhythm and Heart Failure (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: A V1CAMI 2010
Record Dates: First submitted 2015-06-30; First posted 2015-07-08 (Estimated); Last update posted 2015-07-08 (Estimated); Status verified 2015-07

CONDITIONS: Myocardial Infarction
MeSH Terms: conditions — Myocardial Infarction

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Group 1 (Experimental): Patients with documented myocardial infarction in the 7days prior to enrolment and left ventricular ejection fraction >=40% as assessed by echocardiography within 7 days window after MI,who are not candidate to ICD/CRT/IPG implantation after PCI undergo ILR implantation
  Interventions: Device: PCI; Device: ILR implantation

INTERVENTIONS:
Device: PCI
Device: ILR implantation

SUMMARY:
The trial will inform whether detection of ventricular arrhythmias by means of implantable loop recorder (ILR) can help to predict SCD in the large population of survivors of a myocardial infarction with preserved left ventricular function, EF>40%. This may improve risk stratification in these patients, and can inform on the clinical use of subcutaneous monitors to identify post-infarction populations in need for an intervention to prevent sudden death.

ELIGIBILITY:
Inclusion Criteria

* Informed consent signed
* Documented myocardial infarction in the 7days prior to enrolment
* Age > 18 yrs
* Left ventricular ejection fraction >=40% as assessed by echocardiography within 7 days window after MI.

Exclusion Criteria

* subject is unwilling or unable to comply with the study procedures
* documented ventricular tachycardia or survived cardiac arrest outside of an acute coronary syndrome
* Subject has indications for active implanted cardiac medical device (IPG, ICD, CRT).
* contraindications for implantation of a ICM - Planned CABG procedure

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Actual)
Dates: Start 2011-08; Primary Completion 2015-06 (Actual); Study Completion 2015-06 (Actual)

PRIMARY OUTCOMES:
Cardiac arrest | 24 months
Sustained, nonsustained, symptomatic, asymptomatic ventricular tachycardias | 24 months
Ventricular fibrillation | 24 months
Atrial Fibrillation (symptomatic and asymptomatic) | 24 months
Documented Arrhythmic death without evidence of primary non cardiac cause | 24 months

SECONDARY OUTCOMES:
All Arrhythmic events recorded by ILR | 24 months
Changing in treatment strategy, based on physician decision | 24 months
Invasive procedures for arrhythmia treatment | 24 months
Changing in medical treatment (anticoagulation, antiarrhythmic drugs) | 24 months
CV events | 24 months

CONTACTS AND LOCATIONS:
Locations (1):
- State Research Institute of CIrculation Pathology Novosibirsk, Russian Federation, Novosibirsk, Russia

REFERENCES:
- [Derived] Romanov A, Martinek M, Purerfellner H, Chen S, De Melis M, Grazhdankin I, Ponomarev D, Losik D, Strelnikov A, Shabanov V, Karaskov A, Pokushalov E. Incidence of atrial fibrillation detected by continuous rhythm monitoring after acute myocardial infarction in patients with preserved left ventricular ejection fraction: results of the ARREST study. Europace. 2018 Feb 1;20(2):263-270. doi: 10.1093/europace/euw344. PMID 28069838